CLINICAL TRIAL: NCT03283527
Title: Chemoradioresistance in Prospectively Isolated Cancer Stem Cells in Esophageal Cancer-Organoid: RARE STEM-Organoid
Brief Title: Organoid Based Response Prediction in Esophageal Cancer
Acronym: RARESTEM/Org
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: RARESTEM/Organoid
Record Dates: First submitted 2017-08-28; First posted 2017-09-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Organoid; Esophageal Cancer; Chemoradiation
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Current standard treatment of localized esophageal cancer (EC) with neoadjuvant chemoradiotherapy (nCRT) followed by esophagectomy with curative intent results in 30% complete, 40-60% partial and 20% no-response at pathologic examination. Clinical response of nCRT is usually evaluated with PET-CT. However, response measurements are currently still insufficient in optimizing EC treatment. Proper pre-surgical response prediction may allow individualized treatment with esophagus-preservation in complete responders or switching to an alternative treatment in non-responders. Interestingly, in many tumors, a subset of cells has been found to possess cancer stem cell (CSC) properties with associated signaling as drivers of tumor (re-)growth and therapy resistance. Response of CSC-derived tissue resembling in vitro cultured tumor organoids may reflect patient's tumors sensitivity to therapy.

Objective: To create a patient derived organoid model for EC patients to predict the pathologic tumor response to nCRT in clinical practice. This will allow a more personalized approach in future treatment of locally advanced EC.

Study design: Fresh esophageal tumor material will be collected during diagnostic endoscopic ultrasound (EUS) in participating patients. These biopsies will be used to select cancer stem cells, which will be cultured to derive organoids (esophageal cancer patient derived organoids; EC-PDO). When the EC-PDO contain sufficient cells, these cells will be treated with radiotherapy and/or chemotherapy in order to obtain dose-response curves. The response of these EC-PDOs will be compared to the actual tumor response to nCRT treatment in these EC patients, which will be assessed at the definitive pathologic examination of the resection specimen after esophagectomy with curative intent.

Study population: All patients with curatively treatable and resectable esophageal cancer (adenocarcinoma or squamous cell carcinoma) can be included in this trial.

Main study parameters/endpoints: The main endpoint is response prediction to chemoradiotherapy by EC-PDO; the steepness of the dose response survival curve in the organoids in relation to the pathologic response after resection in the clinical situation.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The patients will be asked to undergo 3 to 6 additional biopsies during endoscopic ultrasonography (EUS) for the TNM staging of the tumor. The risk of these additional biopsies is not greater than the biopsies for the diagnosis of EC. The patient will not benefit from participation in this trial.

For the future approach we can get more insight into the mechanism of (chemo)radiation response or resistance to nCRT, which might lead to a better patient selection and more individualized esophageal cancer treatment in the future. This improvement in selection and treatment can result in less over or under-treatment of these EC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adeno- or squamous cell carcinoma of the esophagus
* Age ≥ 18 years
* Candidates for curative treatment; clinical stage T1N+/T2-4aN0-3M0
* Scheduled for endoscopic ultrasound (EUS) procedure for staging and/or treatment purposes
* Written informed consent

Exclusion Criteria:

* Patients who are medically unfit for a curative treatment
* Signs of distant metastases (M1)
* Patients who are mentally disabled or incapable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with histologically proven adenocarcinoma or squamous cell carcinoma of the esophagus, who are candidates for nCRT followed by resection, can be included in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Response prediction by EC-PDO | january 2020
  The main endpoint is response prediction by EC-PDO; the steepness of the dose response survival curve in relation to the pathologic response after resection.

SECONDARY OUTCOMES:
EC-PDO growth rate in-vivo | December 2018- febr 2019
Stem cell characterization measured by the amount of CD24-/CD44+ | March 2018
Radio/Chemo-sensitivity/resistance; the effective dose 50% (ED50%) of CSCs enriched subpopulation will be compared with the ED50% esophageal cancer cell lines. | december 2019/january 2020
Clinical response: based on PET-CT (standard): complete, partial or no response | December 2019/January 2020
Disease free survival (DFS) in months in patients | December 2020/January 2021
Overall survival (OS) in months | December 2020/January 2021

CONTACTS AND LOCATIONS:
Overall Officials: Kristel Muijs, Dr., Principal Investigator — Radiotherapy
Locations (3):
- Netherlands (3):
  - University Medical Center Groningen (UMCG), Groningen
  - Martini Ziekenhuis, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden

IPD SHARING:
Plan to Share IPD: Undecided